CLINICAL TRIAL: NCT01563289
Title: A Randomised, Multicentre, Two-arm, Parallel Group, Double-blind, Placebo-controlled, Comparative Efficacy and Safety Clinical Study of Ibuprofen in Patients With Pain Related to Uncomplicated Ankle Injuries
Brief Title: Efficacy and Safety of Ibuprofen in Patients With Ankle Injuries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0028021; 2011-004496-37 (EudraCT Number)
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2012-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Ibuprofen (Experimental)
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — 3 times a day
  Arms: Ibuprofen
Drug: Placebo — 3 times a day
  Arms: placebo

SUMMARY:
The objective of the study is to evaluate the efficacy and safety of Ibuprofen in patients with ankle injuries.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the efficacy and safety of Ibuprofen versus placebo in patients for the treatment of pain related to uncomplicated ankle injuries.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained.
2. Male and female patients, age in the range of 18-45 years (inclusive).
3. Patients with pain related to uncomplicated ankle injuries (in case of doubt whether it is complicated an X-ray should be taken).
4. Pain related to ankle injuries is scored as moderate or severe by the patient and the injury is less than 24 hours old.
5. Patients with normal or clinically non-significant findings as determined by baseline history, physical examination and vital signs (blood pressure, heart rate and axillary temperature).
6. Comprehension of the nature and purpose of the study and compliance with the protocol requirements.
7. Negative urine pregnancy test (for females only).

Exclusion Criteria:

1. Known hypersensitivity to aspirin or any non-steroidal anti-inflammatory drugs (NSAID).
2. Known history of asthma.
3. Known history of gastric or peptic ulcer or bleeding.
4. Known history of malignancy or other serious diseases.
5. Known history of skin allergy.
6. Known history of cardiac, renal or hepatic insufficiency.
7. Presence of bruises or rash on the skin of ankle.
8. Presence of skin lesions like eczema or psoriasis.
9. Arthritis in the same joint.
10. Alcohol use during the study period or within 48 hours before the study enrolment.
11. Patients judged unable to use the VAS for pain reliably
12. Locally applied NSAID to the painful region/area of study or oral use of NSAID or other analgesics 48 hours before the study enrolment.
13. Other pain killers than rescue medication to be taken during the study.
14. Recurrent sprain at the same joint during the last 6 months.
15. Anticoagulant therapy.
16. Physiotherapy during study period.
17. Open wounds, infected skin or fracture.
18. Any other condition that in the opinion of the investigator would interfere with the evaluation of the results or constitute a health risk for the patient.
19. Pregnant or lactating females.
20. Participation in a drug or device study within 90 days before the study enrolment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Efficacy: visual analog scale (VAS) | Day 7
  VAS pain score change over time from baseline to day 7

SECONDARY OUTCOMES:
Efficacy: VAS | Day 3 and Day 7
  Percentage VAS pain score change from baseline separately to day 3 and 7

CONTACTS AND LOCATIONS:
Overall Officials: Juha-Pekka Kaukonen, MD, Principal Investigator — Terveystalo Lahti
Locations (1):
- Terveystalo Lahti, Lahti, Finland